CLINICAL TRIAL: NCT05143437
Title: Love Together, Parent Together (L2P2): A Feasibility Study of an Ultra-brief Couples Conflict Program for Parents of Young Children
Brief Title: Love Together, Parent Together: A Feasibility Study
Acronym: L2P2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: University of Toronto (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Heather Prime, Assistant Professor, York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: e2021-266
Record Dates: First submitted 2021-11-02; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Family Conflict; Internet-Based Intervention
Keywords: Couples' relationships; Family Systems; Writing Intervention; Non-randomised; Feasibility study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Writing Intervention (Experimental): Couples will take part in three 7-minute online writing sessions over the course of four weeks.
  Interventions: Behavioral: Love Together Parent Together

INTERVENTIONS:
Behavioral: Love Together Parent Together — A brief, low-intensity writing intervention adapted for parents of young children, designed to reduce conflict-related distress, prevent relationship deterioration and encourage the use of conflict reappraisal strategies designed to reduce conflict-related distress, etc.
  Other Names: L2P2

SUMMARY:
The COVID-19 pandemic has introduced additional stressors and challenges to couples' relationships, with potential ripple effects across all family subsystems and child adjustment. Among those who are particularly vulnerable to heightened conflict and lower relationship satisfaction during this time are couples with young children, whose relationships may have already been tenuous prior to the pandemic. The Love Together Parent Together (L2P2) program is a brief, low-intensity writing intervention adapted for parents of young children, designed to reduce conflict-related distress and prevent relationship deterioration. Based on an original writing program by Finkel and colleagues, adaptations include intervention duration and study population. The current study will examine key feasibility metrics related to this adapted intervention program with the goal of identifying problems and informing parameters of future pilot and/or main randomized controlled trials (RCT). The current study is a non-randomised feasibility study, using a single-arm, pre-test/post-test design to primarily assess the feasibility of a large trial, and secondarily to assess the potential effects on outcomes to be used in a future RCT. Couples will be recruited through three community-based agencies with the goal of obtaining a socio-demographically diverse sample. The first 20 couples to enroll will be included. Baseline and post-intervention surveys will be conducted, and a writing intervention will take place (three 7-minute sessions over the course of four weeks). The primary feasibility metrics will include recruitment rates, appropriateness of eligibility criteria, sample diversity, retention, uptake, and adherence, and acceptability. In addition, the researchers will develop an objective primary outcome measure of couple "we-ness" based on analysis of writing samples. The secondary outcomes will include couples' measures (i.e., relationship quality, perceived partner responsiveness, self-reported partner responsiveness, conflict-related distress), and other family outcomes (i.e., parent-child relations, parental/child mental health, and parenting practices). Criteria for success are outlined and failure to meet criteria will result in adaptations to measurement schedule, intervention design, recruitment approaches, and/or other elements of the study design. This feasibility study will inform several components of the procedures used for a subsequent pilot RCT, which will examine the feasibility of the methodology used to evaluate the program (e.g., randomization, attrition to follow up assessment/across groups, and sample size estimation, preliminary effectiveness), and a main trial, which will investigate the effectiveness of the intervention on primary outcome measures as well as mediating pathways.

DETAILED DESCRIPTION:
See attached protocol.

ELIGIBILITY:
Inclusion Criteria:

* Both participants endorse being in a relationship
* Both partners reside in the same home
* There are one or more children under the age of 6 living at home
* Both participants are over age 18 years
* Both members of a couple agree to participate

Exclusion Criteria:

• No current plans or history of separation or divorce as this is meant to be a secondary preventative intervention for couples experiencing some but not severe relationship difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Participants Accessed Per Week | Week 0
  Number of participants accessed (I.e., initiate registration) per week, stratified by recruitment source.
Couple "we-ness" | Week 1-5
  Assessing couple "we-ness" using a content analysis of writing samples collected during the intervention.
Appropriateness of Eligibility Criteria | Week 0
  Percentage of interested participants that meet inclusion criteria (with reasons for exclusion).
Participant Income | Week 0
  The percentage of participants income that is less than or equal to the regional median.
Retention | Week 6
  The percentage of participants who remain in study until the end of the post-intervention assessment.
Uptake | Week 3-5
  The percentage of participants reporting some use of conflict reappraisal outside of sessions.
Adherence | Week 1-5
  The percentage of participants who complete 2/3 intervention sessions.
Acceptability | Week 6
  Looking for the percentage of participants reporting at least 'good' on 80 % or more indicators on an Implementation Acceptability Scale that will assess attitude, burden, perceived effectiveness, and ethicality. Minimum score=7, maximum score=35. Higher scores correspond to better outcomes.
Participants Enrolled Per Week | Week 0
  Number of participants enrolled per week, stratified by recruitment source.
Participant Education | Week 0
  The percentage of participants with less than or equal to a high school degree.
Racial Diversity | Week 0
  The percentage of participants who are a racial minority.
Immigrant Status | Week 0
  The percentage of participants who are an immigrant.
Sexual Diversity | Week 0
  The percentage of participants who are gender and/or sexually diverse.
Risk for Relationship Distress - Dyadic Adjustment | Week 0
  The percentage of participants scoring in the 'clinical' range (>13) on the Dyadic Adjustment Scale. Minimum score=1, maximum score=22. Higher scores correspond to worse outcomes.
Risk for Relationship Distress - COVID-19 Family Stressors | Week 0
  The percentage of participants scoring 'high' (>29) on the COVID-19 Family Stressor Scale. Minimum score=16, maximum score=48. Higher scores correspond to worse outcomes.

SECONDARY OUTCOMES:
Pre-Post Change in Parent Mental Health | Pre-post change from week 0 to week 6.
  Using the Kessler Psychological Distress Scale. Minimum score=10, maximum score=50. Higher scores correspond to worse outcomes.
Pre-Post Change in Parent-Child Relations | Pre-post change from week 0 to week 6.
  Using the Parenting Practices Scale from the Ontario Child Health Study. Minimum score=11, maximum score=55. Higher scores correspond to better outcomes.
Pre-Post Change in Couples' Relationship Quality | Pre-post change from week 0 to week 6.
  Using the Perceived Relationship Quality Scale. Minimum score= 18, maximum score=126. Higher scores correspond to better outcomes.
Pre-Post Change in Conflict-Related Negativity | Pre-post change from week 0 to week 6.
  Using two items following fact-based summary: "I was angry at my partner for his/her behaviour during this conflict," "My partner's behaviour during this conflict was highly upsetting to me". Minimum score=2, maximum score=14. Higher scores correspond to worse outcomes.
Pre-Post Change in Perceived Partner Responsiveness | Pre-post change from week 0 to week 6.
  Using the Perceived Partner Responsiveness-Insensitivity Scale (PRI-R) - Brief Version. Minimum score=8, maximum score=40. Higher scores correspond to better outcomes.
Pre-Post Change in Child Emotional and Behavioural Problems | Pre-post change from week 0 to week 6.
  Scores will be standardized within each age group and used as a single outcome variable.
  Using the Pediatric Symptom Checklist (Baby, Preschool, and Standard versions). The Baby Pediatric Symptom Checklist: Minimum score=0, maximum score=26. Higher scores correspond to worse outcomes.
  The Preschool Pediatric Symptom Checklist (PPSC-17): Minimum score=0, maximum score=36. Higher scores correspond to worse outcomes.
  The Pediatric Symptom Checklist-17: Minimum score=0, maximum score=34. Higher scores correspond to worse outcomes.
Pre-Post Change in Responsiveness Towards Partner | Pre-post change from week 0 to week 6.
  Using the Perceived Partner Responsiveness-Insensitivity Scale (PRI) - Brief with items flipped to reflect responsiveness towards partner. Minimum score=8, maximum score=40. Higher scores correspond to better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Prime, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prime H, Muise A, Benyamin V, Thabane L, Wade M. Love Together, Parent Together (L2P2): a protocol for a feasibility study of a conflict reappraisal writing intervention for interparental couples with young children. Pilot Feasibility Stud. 2022 Aug 6;8(1):170. doi: 10.1186/s40814-022-01115-y. PMID 35933434

DOCUMENTS (2):
  • Study Protocol (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT05143437/Prot_000.pdf
  • Informed Consent Form (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT05143437/ICF_001.pdf